CLINICAL TRIAL: NCT00611845
Title: Aprotinin US Special Access Protocol: An Open Label, Non-Comparative Treatment Protocol for the Use of Aprotinin in Patients Undergoing Coronary Artery Bypass Graft Surgery Requiring Cardiopulmonary Bypass Who Are at Increased Risk of Blood Loss and Transfusion
Brief Title: Aprotinin US Special Access Protocol
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Other Study IDs: 13087
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Hemorrhage
Keywords: CABG surgery requiring CPB and at increased risk of bleeding and blood transfusion
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Aprotinin

INTERVENTIONS:
Drug: Aprotinin (Trasylol, BAYA0128) — Trasylol at either 1,000,000 KIU or 2,000,000 KIU

SUMMARY:
This is a special access protocol that will allow physicians access to aprotinin during the temporary marketing suspension. The program will provide aprotinin for treatment of surgical patients undergoing coronary artery bypass graft (CABG) surgery requiring cardiopulmonary bypass (CPB) who are at increased risk of bleeding and transfusion when, in the opinion of the treating physician, the patients require it, there is no acceptable alternative therapy, and when there is a clearly favorable benefit-risk for the drug in that individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients undergoing cardiopulmonary bypass in the course of coronary artery bypass graft surgery who are at an increased risk for blood loss and blood transfusion. These patients may include the following:

  * Patients receiving preoperative antithrombotic drugs (e.g., clopidogrel, aspirin),
  * Patients undergoing repeat CABG or complex CABG procedures,
  * Patients undergoing urgent or emergent CABG procedures,
  * Patients who refuse to receive allogeneic blood products for religious or other reasons,
  * Patients undergoing primary CABG with advanced age or multiple comorbidities such as preoperative anemia, coagulopathies, diabetes mellitus, and peripheral vascular disease
* The physician has determined that no acceptable alternative comparable therapy is available for the patient and that there is a clearly favorable benefit-risk for the drug in that individual patient
* Documented, signed, dated informed consent obtained prior to entry into the study

Exclusion Criteria:

* Patients with a known or suspected previous aprotinin exposure during the last 12 months. Aprotinin may also be a component of some fibrin sealant products, and the use of these products should be considered when evaluating previous aprotinin exposure
* Patients with a known or suspected allergy to aprotinin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (16):
  - Decatur, Alabama
  - Glendale, California
  - Pismo Beach, California
  - Santa Monica, California
  - Ventura, California
  - Fort Wayne, Indiana
  - Edgewood, Kentucky
  - New Brunswick, New Jersey
  - Asheville, North Carolina
  - Medford, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Knoxville, Tennessee
  - Lynchburg, Virginia
  - Milwaukee, Wisconsin
  - Wausau, Wisconsin